CLINICAL TRIAL: NCT05158608
Title: A Randomized, Open-label, Single-center Study Comparing Cyclophosphamide at a Dose of 25 mg/kg/Day and Cyclophosphamide at a Dose of 50 mg/kg/Day in Graft Versus Host Disease Prophylaxis
Brief Title: Comparison of PT-Cy at a Dose of 25 mg/kg/Day and PT-Cy at a Dose of 50 mg/kg/Day in GVHD Prophylaxis
Acronym: CY25
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Mikhail Drokov, MD, PhD, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CY25
Record Dates: First submitted 2021-12-12; First posted 2021-12-15 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Graft Versus Host Disease; Hematologic Malignancy; Cyclophosphamide Adverse Reaction
Keywords: Allogeneic transplantation; Graft-versus-host-disease prophylaxis; Post-transplant cyclophosphamide
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Cyclophosphamide; trihexyltetradecylphosphonium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide on day +3,+4 at dose 50 mg/kg/day (Active Comparator): Post-transplantation Cyclophosphamide will be apply for GVHD prophylaxis on day +3,+4 at dose 50 mg/kg/day in combination with cyclosporine A at 3 mg/kg/day from day +5 and mycophenolate mofetil at dose 30-45mg/kg/day from day +5.
  Interventions: Drug: Post-transplantation Cyclophosphamide at dose 50 mg/kg/day
- Cyclophosphamide on day +3,+4 at dose 25 mg/kg/day (Experimental): Post-transplantation Cyclophosphamide will be apply for GVHD prophylaxis on day +3,+4 at dose 25 mg/kg/day in combination with cyclosporine A at 3 mg/kg/day from day +5 and mycophenolate mofetil at dose 30-45mg/kg/day from day +5.
  Interventions: Drug: Post-transplantation Cyclophosphamide at dose 25 mg/kg/day

INTERVENTIONS:
Drug: Post-transplantation Cyclophosphamide at dose 25 mg/kg/day — Post-transplantation Cyclophosphamide will be apply for GVHD prophylaxis on day +3,+4 at dose 25 mg/kg/day in combination with cyclosporine A at 3 mg/kg/day from day +5 and mycophenolate mofetil at dose 30-45mg/kg/day from day +5.
  Other Names: Endoxan; Cyphos
  Arms: Cyclophosphamide on day +3,+4 at dose 25 mg/kg/day
Drug: Post-transplantation Cyclophosphamide at dose 50 mg/kg/day — Post-transplantation Cyclophosphamide will be apply for GVHD prophylaxis on day +3,+4 at dose 50 mg/kg/day in combination with cyclosporine A at 3 mg/kg/day from day +5 and mycophenolate mofetil at dose 30-45mg/kg/day from day +5.
  Other Names: Endoxan; Cyphos
  Arms: Cyclophosphamide on day +3,+4 at dose 50 mg/kg/day

SUMMARY:
This is a two arm open label phase III clinical trial. Adult patients with hematological malignancies undergoing allogeneic HSCT from any donor are eligible for the study if they meet the standard criteria defined in the investigator's institutional standard operation procedures (SOPs), meet all inclusion criteria, and do not satisfy any exclusion criteria. Patients will receive reduced-intensity conditioning regimen of fludarabine, busulfan (treosulfan). Patients will receive PTCy at different dose (25 mg/kg/day vs 50 mg/kg/day on day +3,+4 in combination with calcineurin inhibitors and mofetil mycophenolate) as GvHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an indication for allogeneic hematopoietic stem cell transplantation

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute graft-versus-host disease, grades II-IV | 180 days
  MAGIC criteria
Incidence of chronic GVHD, moderate and severe (NIH criteria) | 365 days
  NIH criteria

SECONDARY OUTCOMES:
Overall survival analysis | 365 days
  Kaplan-Meier survival analysis
Event-free survival analysis | 365 days
  Kaplan-Meier survival analysis
Non-relapse mortality analysis | 365 days
  Kaplan-Meier survival analysis, competing risk analysis
Incidence of graft failure and poor graft function | 365 days
  Kaplan-Meier survival analysis, competing risk analysis
Incidence of 30-Day Readmission | 365 days
  Kaplan-Meier survival analysis, competing risk analysis

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnikova, MD, D.Sc, Principal Investigator — National Research Center for Hematology